CLINICAL TRIAL: NCT00278538
Title: Cyclophosphamide and rATG/Rituximab in Patients With Systemic Lupus Erythematosus: Phase II Trial
Brief Title: Cyclophosphamide and Rabbit Antithymocyte Globulin (rATG)/Rituximab in Patients With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DI SLE.Auto2003
Record Dates: First submitted 2006-01-15; First posted 2006-01-18 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2019-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Stem cell, Autoimmune disease, Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hematopoietic Stem Cell Transplant Regimen 2 (Experimental): Autologous Hematopoietic Stem Cell Transplantation: Rituximab, rATG and Cyclophosphamide regimen
  Interventions: Biological: Hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: Hematopoietic stem cell transplantation — Autologous hematopoietic stem cell transplantation

SUMMARY:
This study is designed to examine whether treating patients with lupus with high dose cyclophosphamide together with rATG/rituximab (drugs which reduce the function of the immune system), followed by return of their previously collected stem cells will result in improvement in the disease. Stem cells are undeveloped cells that have the capacity to grow into mature blood cells, which normally circulate in the blood stream. The purpose of the intense chemotherapy is to destroy the cells in the immune system which may be causing this disease. The purpose of the stem cell infusion is to produce a normal immune system that will no longer attack body. The study purpose is to examine whether this treatment will result in improvement in the lupus disease.

DETAILED DESCRIPTION:
Mobilization Participants will be administered Cyclophosphamide at 2.0 g/m2 in 200 ml of normal saline (NS) over 1 hour. Hydration with 0.9 NS at approximately 100-250-ml/ hour will begin 4 hours prior to cyclophosphamide and continued for 24 hours after termination of cyclophosphamide. Urine output approximately greater than 100 ml/hour should be maintained.

Granulocyte-colony stimulating factor (G-CSF) will be administered subcutaneously at 5-10 mcg/kg/day and will be started 5 days after termination of cyclophosphamide administration.

After the absolute neutrophil count is greater than 1000/ul or after hematological nadir, leukapheresis using a continuous flow blood cell separator will be initiated. A 10-15 liter apheresis will be performed unless stopped earlier for clinical judgment of toxicity (e.g., numbness, tetany). The G-CSF will continue until apheresis is discontinued. If necessary, platelets will be transfused to greater than 60,000/ul prior to each apheresis.

Conditioning Regimen Mesna: 50mg/kg/day x 4 days will be given intravenously over 24 hours.

Cyclophosphamide: 50 mg/kg/day x 4 days (the lesser of ideal or actual weight) will be given intravenously over 1 hour in 250 cc of normal saline on days -5 through -2.

Hydration: approximately 50-200cc/hour in adults should begin 6 hours before cyclophosphamide and continue until 24 hours after the last cyclophosphamide dose. Hydration rates need to be individually adjusted by daily weights to maintain dry weight count. Twice daily weights will be obtained. Warning: Participants with renal insufficiency are prone to volume overload. Early institution of ultrafiltration or dialysis is recommended.

rATG 0.5mg/kg will be given IV on day -5, 1.0mg/kg will be given on day

-4, 1.5mg/kg will be given IV on days -3, -2, -1 (no dose adjustment). It will be given over 10 hours. Premedicate with Solumedrol 250mg IV, acetaminophen 650mg po qd and diphenhydramine 25mg 30 minutes before infusion.

Rituximab 500mg/day will be given IV on days -6 and +1. At the first dose (D-6), rituximab infusion will be started at 50mg/h and escalate the infusion rate by 50mg every 30minutes to a maximum of 400mg/h. Starting the second dose (days -4, -2 and +1). IV infusion will be started at 100mg/h and escalate the infusion rate 100mg every 30minutes to a maximum of 400mg/h. Premedicate with Solumedrol 250mg IV, acetaminophen 650mg po qd and diphenhydramine 25mg 30 minutes before infusion on days -6 and +1. Premedicate acetaminophen 650mg po qd and diphenhydramine 25mg 30 minutes before infusion on days -4 and -2.

Stem Cell Reinfusion Previously collected stem cells will be reinfused on day 0 as noted in Table 4. The stem cells are infused over approximately 20 minutes through the central venous catheter, such as a peripherally inserted central catheter (PICC line). Following stem cell reinfusion, routine daily labs will be obtained including complete blood count (CBC), chemistry panel, and liver function tests. Antibiotics and blood transfusions will be administered as required by clinical judgment.

ELIGIBILITY:
Inclusion Criteria:

* Ages 15 to 60 years old
* Meet at least 4 of 11 American College of Rheumatology (ACR) Classification criteria for systemic lupus erythematosus (SLE) (see Appendix 16.2)
* Meet one of following five:

  1. For lupus nephritis, participants must fail pulse cyclophosphamide (500 to 1000 mg/m2 monthly for a minimum of 6 months). Failure is defined as meeting criteria to be considered as BILAG renal category A.
  2. For visceral organ involvement other than nephritis, participants must be BILAG cardiovascular/respiratory category A, vasculitis category A, or neurologic category A and must fail at least 3 months of oral or IV cyclophosphamide and be corticosteroid dependent. Steroid dependence being defined as at least 3 months of steroid therapy and inability to wean corticosteroid to less than 20 mg/day of prednisone or equivalent.
  3. For cytopenias that are immune mediated, participants must be BILAG hematologic category A. Participants must fail corticosteroids (either oral prednisone > 0.5 mg/kg/day for more than 6 months or pulse methylprednisolone for at least one cycle of three days), and at least one of the following: azathioprine at 2 mg/kg/day for at least 3 months, mycophenolate mofetil 2 grams daily for more than 3 months, cyclophosphamide intravenously or orally for at least 3 months, or cyclosporine at least 3 mg/kg/day for at least 3 months, danazol for at least 3 months, or splenectomy.
  4. For mucocutaneous disease, participants must meet BILAG mucocutaneous category A, be unable to be weaned from prednisone to less than 0.5 mg/kg/day for more than 6 months and obvious cushingoid habitus, and have received at least one of the following: azathioprine at 2 mg/kg/day for at least 3 months, methotrexate at 15mg/week for at least 3 months, cyclophosphamide intravenously or orally for at least 3 months, or cyclosporine at least 3 mg/kg/day for at least 3 months.
  5. For arthritis/myositis, participants must meet BILAG musculoskeletal category A, be unable to be weaned from prednisone to less than 0.5 mg/kg/day for more than 6 months and obvious cushingoid habitus, and have received at least one of the following: azathioprine at 2 mg/kg/day for at least 3 months, methotrexate at 15mg/ week for at least 3 months, cyclophosphamide intravenously or orally for at least 3 months, or cyclosporine at least 3 mg/kg/day for at least 3 months.
* Able to give informed consent.
* If indication for hematopoietic stem cell transplant (HSCT) is nephritis, a renal biopsy must demonstrate the potential of a reversible (non-fibrotic) component indicating that if successful the participant would not be likely to be permanently dialysis-dependent after transplant.
* Since the BILAG is only one of multiple indices for SLE, patients may also be candidates if despite prior immune suppression therapy as described above, patients are still on active immune suppression (more than 10mg a day of prednisone).
* Patients with SLE whose major manifestation is Antiphospholipid syndrome (APS) may be candidates without prior immune suppression therapy if they have had a visceral organ thrombotic or embolic event despite anticoagulation.
* Patients with SLE whose major manifestation is Antiphospholipid syndrome (APS) may be candidates without prior immune suppression therapy if they have had a visceral organ thrombotic or embolic event despite anticoagulation.

Exclusion Criteria:

* HIV positive
* Ongoing malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the participant is judged to be cured by local surgical therapy, such as head and neck cancer, or stage I or II breast cancer will be considered on an individual basis by the investigators doing the final screening for participant qualification.
* Positive pregnancy test, inability or unwillingness to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
* Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
* Diffusing capacity of lung for carbon monoxide (DLCO) < 45% of predicted unless attributed to active lupus.
* Resting left ventricular ejection fraction (LVEF) < 40% unless attributed to active lupus.
* Known hypersensitivity to E Coli derived proteins.
* Transaminases greater than 2 times normal unless attributed to active lupus.
* Positive tuberculosis skin test
* Any active infection
* Any co-morbid illness that in the opinion of the investigator would jeopardize the ability of the subject to tolerate the study.
* Failure to collect at least 2.0 x 106 cluster of differentiation 34 (CD34+) cells/kg
* Antinuclear antibody (ANA)-negative

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2005-09-23 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Northwestern University, Chicago, Illinois

REFERENCES:
- [Background] Burt RK, Han X, Gozdziak P, Yaung K, Morgan A, Clendenan AM, Henry J, Calvario MA, Datta SK, Helenowski I, Schroeder J. Five year follow-up after autologous peripheral blood hematopoietic stem cell transplantation for refractory, chronic, corticosteroid-dependent systemic lupus erythematosus: effect of conditioning regimen on outcome. Bone Marrow Transplant. 2018 Jun;53(6):692-700. doi: 10.1038/s41409-018-0173-x. Epub 2018 May 31. PMID 29855561
- [Derived] Burt RK, Craig RM, Milanetti F, Quigley K, Gozdziak P, Bucha J, Testori A, Halverson A, Verda L, de Villiers WJ, Jovanovic B, Oyama Y. Autologous nonmyeloablative hematopoietic stem cell transplantation in patients with severe anti-TNF refractory Crohn disease: long-term follow-up. Blood. 2010 Dec 23;116(26):6123-32. doi: 10.1182/blood-2010-06-292391. Epub 2010 Sep 13. PMID 20837778
- See also: Bone Marrow Transplant — https://www.nature.com/articles/s41409-018-0173-x

RESULTS

PARTICIPANT FLOW:
Groups:
- Hematopoietic Stem Cell Transplantation: Autologous hematopoietic stem cell transplantation will be performed
  Hematopoietic stem cell transplantation: Autologous hematopoietic stem cell transplantation
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplantation
Started | 32
Completed | 30
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 32 [16 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: The primary efficacy outcome is overall survival.
Time Frame: 6 months, then yearly x 5 years after transplant
Population: The # analyzed at 6 mos.- 4 years differs from the overall participant # analyzed because 2 participants were declined HSCT due to comorbidities and 2 died within 6 mos. after HSCT unrelated to the treatment. The # analyzed at 5 years differs from the overall participants analyzed due to an unrelated treatment death at 4 years after HSCT.
  .
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 30
Participants
  6 Month Post Transplant Survival: Total Participant Survival | 28
  6 Month Post Transplant Survival: Non Treatment Related Death | 2
  1 Year Post Transplant Survival: number analyzed (Participants) | 28
  1 Year Post Transplant Survival: Total Participant Survival | 28
  1 Year Post Transplant Survival: Non Treatment Related Death | 0
  2 Year Post Transplant Survival: number analyzed (Participants) | 28
  2 Year Post Transplant Survival: Total Participant Survival | 28
  2 Year Post Transplant Survival: Non Treatment Related Death | 0
  3 Year Post Transplant Survival: number analyzed (Participants) | 28
  3 Year Post Transplant Survival: Total Participant Survival | 28
  3 Year Post Transplant Survival: Non Treatment Related Death | 0
  4 Year Post Transplant Survival: number analyzed (Participants) | 28
  4 Year Post Transplant Survival: Total Participant Survival | 27
  4 Year Post Transplant Survival: Non Treatment Related Death | 1
  5 Year Post Transplant Survival: number analyzed (Participants) | 27
  5 Year Post Transplant Survival: Total Participant Survival | 27
  5 Year Post Transplant Survival: Non Treatment Related Death | 0

ADVERSE EVENTS:
Time Frame: 5 year
Arm/Group | Hematopoietic Stem Cell Transplantation
All-Cause Mortality (participants affected / at risk) | 3/30
Serious Adverse Events (participants affected / at risk) | 5/30
Other Adverse Events (participants affected / at risk) | 10/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=30)
Elevated Troponin (Cardiac disorders) | 1 (1) — Grade 4 Toxicity During HSCT Hospitalization
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) — Grade 4 Toxicity During HSCT Hospitalization
Intracranial Hemorrhage (General disorders) | 1 (1) — Grade 4 Toxicity During HSCT Hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=30)
Neutropenic Fevers (Infections and infestations) | 10 (10) — Grade 3 Toxicity During HSCT Hospitalization
Hypokalemia (Metabolism and nutrition disorders) | 8 (8) — Grade 3 Toxicity During HSCT Hospitalization
Hypertension (Cardiac disorders) | 7 (7) — Grade 3 Toxicity During HSCT Hospitalization
Hyperglycemia (Metabolism and nutrition disorders) | 6 (6) — Grade 3 Toxicity During HSCT Hospitalization
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (5) — Grade 3 Toxicity During HSCT Hospitalization
Dyspnea (General disorders) | 5 (5) — Grade 3 Toxicity During HSCT Hospitalization
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3) — Grade 3 Toxicity During HSCT Hospitalization
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) — Grade 3 Toxicity During HSCT Hospitalization
Elevated Transaminase (General disorders) | 2 (2) — Grade 3 Toxicity During HSCT Hospitalization
Chest Pain (Cardiac disorders) | 2 (2) — Grade 3 Toxicity During HSCT Hospitalization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-10-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT00278538/Prot_000.pdf
  • Statistical Analysis Plan (2015-10-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT00278538/SAP_001.pdf